CLINICAL TRIAL: NCT03951545
Title: Clinical and Radiological Impact of Tibial Cutting Int Total Knee Arthroplasty, Accelerated Navigation Versus Extramedullary Targeting : a Randomized Prospective Study
Brief Title: Clinical and Radiological Impact of Tibial Cutting Int Total Knee Arthroplasty, Accelerated Navigation Versus Extramedullary Targeting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: PO18142
Record Dates: First submitted 2018-11-07; First posted 2019-05-15 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2018-12

CONDITIONS: Gonarthrosis
Keywords: Osteoarthritis Knee; Knee prosthesis; Patient satisfaction
MeSH Terms: conditions — Osteoarthritis, Knee; Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mechanical group (Active Comparator): Group of patients whose tibial sections will be performed using extramedullary mechanical sighting
  Interventions: Procedure: First line total knee replacement for gonarthrosis .
- Gyroscopic group (Experimental): Group whose tibial sections will be performed using gyroscopic and accelerometric navigation (I-Assist) will be randomized
  Interventions: Procedure: First line total knee replacement for gonarthrosis .

INTERVENTIONS:
Procedure: First line total knee replacement for gonarthrosis . — Patients requiring 1st line total knee replacement for gonarthrosis with a Hip knee angle (HKA) between 170° and 183°. In the first group (Mechanical) the total knee replacement will be performed with a tibial cut by using extramedullary mechanical sighting and in the second group (Gyroscopic) by using gyroscopic and accelerometric navigation (I-Assist).

SUMMARY:
Type of study :

Superiority study, comparative, randomized, double-blind (patient and evaluator will be blind from the randomization group), multicenter, prospective inclusion. Two groups of patients will be compared: a group of patients whose tibial sections will be performed using extramedullary mechanical sighting and a group whose tibial sections will be performed using gyroscopic and accelerometric navigation (I-Assist) will be randomized. Randomization will be performed with a 1/1 ratio per block.

Population :

Patients requiring 1st line total knee replacement for gonarthrosis with a Hip knee angle (HKA) between 170° and 183° who have agreed to participate in the study. Patients who have already undergone surgery on the same knee (uni-compartmental prosthesis, total knee replacement, tibial or femoral osteotomy for re-alignment, with the exception of arthroscopy) or who have vicious calls will not be included in the study.

The number of subjects required was calculated using NQUERY 4.0 software for the main endpoint data, with the following assumptions: 51% of patients reaching the tibial cut target angles for the "extramedullary mechanical aiming" technique and 68% of patients reaching the tibial cut target angles for the I-Assist gyroscopic and accelerometric navigation technique. With an alpha risk of 5%, a power of 90%, and bilateral test, the number was estimated at 174 per group. Taking into account a percentage of included patients for whom total knee arthroplasty will not be performed of 10%, it is planned to include a total of 382 patients.

Main judgment criteria :

Achievement of the target tibial slope of 3°+/-2° and the target tibial varus/valgus at +/-2°. The tibial slope is defined by the angle (in degrees) between the mechanical axis of the tibia in profile and the tangent to the tibial cut. The varus/valgus tibial is the angle formed between the mechanical axis of the front tibia and the tangent to the tibial cut.

Investigation plan :

Proposal to participate in the research to any eligible patient at the time of a preoperative consultation with the orthopaedic surgeon. If the patient agrees to participate in the research (signature of the informed consent form), a randomization will be performed to determine the group of bone cutting technique. The patient will be blind to the result of randomization.

The clinical follow-up of the patient will not be modified by the study, with as usual:

* A 6-week consultation with interrogation, clinical and radiographic examination (Face and profil x-rays, axial patella views)
* A 3-month consultation with interrogation, clinical and radiographic examination (Face and profil x-rays, axial patella views, telemetry of the lower limbs in charge and full profile leg x-rays).
* Measurements of the radiographic judgement criteria will be performed by two orthopaedic surgeons and a blind radiologist of the cutting technique used. The tibial slope will be analyzed on the entire leg radiograph in profile at 3 months. Coronal alignment will be studied on telemetry of the front lower limbs loaded at 3 months.
* Joint amplitudes and patient satisfaction will be assessed at 3 months postoperatively with the New IKS score, by a blind surgeon of the surgical technique used.

Statistical analysis plan :

* Comparison of the characteristics of the 2 groups
* Analysis of the main endpoint: comparison of the percentage of patients with the target tibial slope achieved in both groups by Chi2 test or an accurate Fisher test, depending on the application conditions.
* Analysis of secondary judgment criteria by Student, Wilconxon, Chi2 or exact Fisher tests, depending on the application conditions.

ELIGIBILITY:
Inclusion Criteria:

* Gonarthrosis
* Hip Knee Angle between 170° and 183°
* Agreed to participate in the study

Exclusion Criteria:

* Already undergone surgery on the same knee:

  * Uni-compartmental prosthesis
  * Total Knee Replacement
  * Tibial or femoral osteotomy for re-alignment
* Vicious calls

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Estimated)
Dates: Start 2018-11-21 (Actual); Primary Completion 2021-02-21 (Estimated); Study Completion 2021-08-21 (Estimated)

PRIMARY OUTCOMES:
Achievement of the target tibial slope and the target tibial varus/valgus | 3 months
  Achievement of the target tibial slope of 3° +/- 2° and the target tibial varus/valgus +/- 2°. The tibial slope is defined by the angle (in degrees) between the mechanical axis of the tibia in profile and the tangent to the tibial cut. The tibial varus/valgus is the angle formed between the mechanical axis of the front tibia and the tangent to the tibial cut. This radiological evaluation is a usual assessment used in the follow-up of patients operated for a total knee replacement.

SECONDARY OUTCOMES:
Achievement of target global coronal alignement | 3 months
  Achievement of the global coronal alignment target +/- 3° defined in the preoperative pase. Coronal alignment is defined by the HKA angle, the angle (in degrees) between the center of the femoral head, the center of the knee and the center of the tibio-fibluar mortise. This radiological evaluation is a usual assessment used in the follow-up of patients operated for a total knee replacement.
Patient satisfaction: New IKS score | 3 months
  Patient satisfaction will be assessed using the New International Knee Society score (New IKS score) collected by a blind investigator.
  The new IKS score was validated in French in 2014 (Debette C, Parratte S, Maucort-Boulch D, Blanc G, Pauly V, Lustig S, Servien E, Neyret P, Argenson JN.
  French adaptation of the new Knee Society Scoring System for total knee arthroplasty. Orthop Traumatol Surg Res. 2014 Sep;100(5):531-4.) New IKS score range from 0 to 200 with a physical score on 100 points (pain, knee' mobility, abnormal laxity, flexion deformity and Hips knee Ankle) and a functional score on 100 points (walking distance, difficulty with stairs and use of walking aids).

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France